CLINICAL TRIAL: NCT00573742
Title: Non-interventional Study on Uncontrolled Hypertensive Patients for Evaluating Efficacy of Candesartan Cilexetil as Monotherapy or add-on Therapy.
Brief Title: Efficacy Observational Study of Candesartan Cilexetil on Hypertensive Patients
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: MC MD, AstraZeneca
Other Study IDs: NIS-CRO-ATA-2007/1
Record Dates: First submitted 2007-12-13; First posted 2007-12-14 (Estimated); Last update posted 2010-08-19 (Estimated); Status verified 2010-08

CONDITIONS: Primary Hypertension
Keywords: hypertension
MeSH Terms: conditions — Essential Hypertension; Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Candesartan Cilexeotil 16mg

SUMMARY:
The purpose of this study is to observe treatment with candesartan cilexetil 16mg for 8 weeks, in uncontrolled hypertensive patients, in improvement of achieving of treatment goals and impact on blood pressure level in patients with uncontrolled hypertension treated with candesartan cilexetil.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of essential hypertension (mild or moderate as defined in European Guidelines of Hypertension, 2003), that are treated already with candesartan cilexetil 16mg o.d. within last 2 weeks or more, according to Romanian approved Atacand SPC. Written informed consent to allow access and use(analysis) of data collected

Exclusion Criteria:

* Patients not to be included in the programme: patients who have any contraindication to the product as detailed in Romanian approved Atacand SPC. Use of specific concomitant medication known to present a potential safety concern according to Romanian approved SPC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hypertensive patients not at BP target (according to ESC Guideline for the management of hypertension, 2003), already treated with candesartan cilexetil 16 mg/day
Sampling Method: Non-Probability Sample
Enrollment: 1940 (Actual)
Dates: Start 2007-09; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mihai Isvoranu, Study Chair — AstraZeneca; Gabriela Teodorescu, Study Director — AstraZeneca
Locations (16):
- Romania (16):
  - Research Site, Bacau
  - Research Site, Brasov
  - Research Site, Brăila
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Constanța
  - Research Site, Craiova
  - Research Site, Galati
  - Research Site, Ghiroda
  - Research Site, Iași
  - Research Site, Lugoj
  - Research Site, Oradea
  - Research Site, Piteşti
  - Research Site, Ploieşti
  - Research Site, Sibiu
  - Research Site, Timișoara